CLINICAL TRIAL: NCT06324084
Title: Pathophysiology of Osteoporosis: Role of Hidden Cortisol Excess and Its Predictors in Bone Fragility (PNRR-MAD-2022-12375951)
Brief Title: PATHophysiology of OSteoporosis: Role of Hidden Cortisol Excess and Its Predictors in Bone Fragility
Acronym: PATHOS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05M201
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Osteoporosis; Bone Fracture; Cortisol Excess
Keywords: Osteoporosis; Cortisol
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum samples for the assessment of bone turnover markers Blood samples for the assessment of circulating microRNAs 24-hour urinary samples for the assessment of 24-hour urinary free cortisol/free cortisone ratio DNA isolated from blood samples for the determination of 11ßHSD1, GR and B2AR gene polymorphisms Fecal samples for the analysis of gut microbiome composition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoporosis is a chronic skeletal disease which leads to a decrease in bone strength which increases the risk of fractures.

Clinically overt hypercortisolism leads to hypertension, central obesity, diabetes and osteoporosis. More recently, even the condition of mild and asymptomatic hypercortisolism has been associated with increased prevalence of chronic complications of cortisol excess and mortality. In patients with osteoporosis this form of hypercortisolism may remain occult (hidden hypercortisolism, HidHyCo).

Although asymptomatic, however, this subtle cortisol excess is associated with an increased risk of osteoporosis and fragility fractures.

Moreover, HidHyCo prevalence seems to be increased in osteoporotic patients. The HidHyCo case finding is of utmost importance. However, given the high prevalence of bone fragility and the relatively low diagnostic accuracy of the currently available tests for the HidHyCo detection, a mass screening for HidHyCo is considered unthinkable. As now, no guidelines are available for addressing the HidHyCo screening in osteoporosis.

Therefore, the aims of the present study are the following: i) to assess the HidHyCo prevalence in a sample of osteoporotic patients; ii) to compare the clinical characteristics between osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo in order to determine the clinical characteristics more frequently associated with the HidHyCo presence and to identify those osteoporotic patients worthy of HidHyCo screening; iii) to further investigate bone quality and turnover in HidHyCo patients, to characterize HidHyco patients from a molecular and genetic point of view and to evaluate the pathogenetic mechanisms explaining the negative effects of endogenous cortisol excess on bone health in these patients and the potential role of the genetic background and of the gut microbiome.

The HidHyCo could be present in a not negligible percentage of osteopenic/osteoporotic patients. In these patients, osteoporosis and, if present, other comorbidities can improve by the surgical resection of the adrenal or pituitary adenoma if feasible, or by the use of drugs able to modulate cortisol secretion or glucocorticoid sensitivity. Moreover, the case-finding could be reserved in those patients at higher risk of having HidHyCo, therefore, reducing the costs of a scarcely specific mass screening.

DETAILED DESCRIPTION:
Clinically overt hypercortisolism leads to hypertension, diabetes and osteoporosis. More recently, even the condition of mild and asymptomatic hypercortisolism has been described to be associated with increased prevalence of chronic complications of cortisol excess and mortality. In patients with osteoporosis this form of hypercortisolism may remain occult (hidden hypercortisolism, HidHyCo).

The HidHyCo prevalence in the general population is estimated to be 0.2-2%, but it has been reported up to 9.9% and 17.6% in patients with low bone mineral density and with fragility fracture, respectively. However, given the high prevalence of bone fragility and the relatively low specificity of the available tests for the HidHyCo detection, screening all osteoporotic patients for HidHyCo is considered unthinkable and no guidelines are available for addressing the HidHyCo screening in osteoporosis.

At present, data regarding the osteoporosis characteristics more frequently associated with HidHyCo have been not reported, even though some data suggest that the coexistence of osteopenia with hypertension treated with at least 2 drugs or with not well controlled hypertension and/or diabetes or with a history of cardiovascular events may increase the probability of HidHyCo.

Moreover, scarce and discordant data are available on the pathogenesis of the bone damage due to a subtle cortisol excess and on the possible role of individual bone sensitivity to cortisol and of microbiome composition.

Therefore, the aims of the current project are the following: i) to assess the prevalence of HidHyCo, ii) to determine the characteristics predictive of the presence of this condition in patients with apparently primary osteoporosis, iii) to evaluate the pathogenetic mechanisms explaining the negative effects of this slight cortisol excess on bone and the potential role of the genetic background and of the gut microbiome.

In all patients who have been included in the study and who have given the informed consent to participate in the study 1 mg overnight dexamethasone suppression test (F-1mgDST) will be performed. In all subjects with F-1mgDST >1.8 mcg/dL, cortisol levels after two-day low dose (2 mg/day) dexamethasone suppression test (F-2mgx2dDST) will be measured.

Patients with F-2mgx2dDST above >1.8 mcg/dL will be considered affected with HidHyCo and will be managed following the available guidelines for hypercortisolism.

The HidHyCo prevalence in osteopenic/osteoporotic patients and its 95% interval confidence will be calculated.

Moreover, in all recruited patients the following vital and anthropometric parameters will be recorded: blood pressure, heart rate, weight, height, body mass index (BMI), abdominal circumference and waist-to-hip ratio. Moreover, the following variables will be collected: familiar history of fragility fracture, smoking habit, main comorbidities, history of falls, previous clinical fragility fractures, ongoing pharmacological treatment (in particular type and number of antihypertensive, lipid lowering, anti-diabetic and anti-osteoporotic drugs), previous anti-osteoporotic treatments, in females regularity of menses or age of menopause and in males testosterone levels. Questionnaires for assessing daily calcium intake and physical activity will be administered to all patients. At the time of enrolment, the results of first tier investigations according to national guidelines (i.e. serum erythrocyte sedimentation rate, complete blood count, serum protein electrophoresis, serum calcium levels, serum phosphate levels, total alkaline phosphatase, serum creatinine, 24-h urinary calcium) will be also registered. Moreover, other calcium-phosphate metabolism parameters (i.e. serum ionized calcium, serum parathyroid hormone, serum 25-OH-vitamin D, serum ß-CrossLaps, bone alkaline phosphatase) and routine determinations (i.e. fasting glucose, insulin, glycated haemoglobin, total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides, transaminases) will be recorded, if available.

According to the good clinical practice, in all patients bone mineral density will be assessed by dual-energy X-ray Absorptiometry (Hologic or Lunar bone densitometers) and the presence of asymptomatic vertebral fractures will be checked by conventional spinal radiographs using the semi-quantitative visual assessment described by Genant et al., defined as a reduction of >20% in anterior, middle, or posterior vertebral height.

The investigators will compare the clinical and biochemical characteristics of osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo. The sample size has been calculated in order to have an adequate number of HidHyCo cases to determine the characteristics of osteoporotic patients suggestive for the presence of HidHyCo. Since HidHyCo may be estimated to have at least a 3% prevalence in osteoporotic patients, a sample of 1500 osteoporotic patients should be adequate to find no less than 45 HidHyCo cases.

To further investigate bone quality and turnover in HidHyCo patients, to characterize HidHyco patients from a molecular and genetic point of view and to evaluate the pathogenetic mechanisms explaining the negative effects of endogenous subtle cortisol excess on bone health and the potential role of the genetic background and of the gut microbiome.

In patients found to be affected with HidHyCo and in age-, sex- and BMI-matched patients without HidHyCo (with a case-control ratio of 1:2) the investigators will:

i) assess bone turnover markers and new potential serum markers of bone status, such as those involved in the Wnt-ßcatenin signaling; ii) perform Radiofrequency echographic multi spectrometry (REMS), a non-ionizing skeleton technique performed employing a new dedicated echographic device (EchoStation, Echolight Spa, Lecce, Italy) to further investigate bone quality characteristics that are not included in DXA-measured BMD, such as the Fragility Score (FS).

iii) assess circulating microRNAs (miRNAs, i.e. small non coding single-stranded RNAs that have emerged as important post transcriptional regulators of gene expression) expression profile; iv) assess cortisol peripheral activation, as expressed by the 24-hour urinary free cortisol/free cortisone ratio (i.e., the higher the R-UFF/UFE, the higher tissues exposure to active glucocorticoids), measured by liquid chromatography-tandem mass spectrometry and its relationship with the polymorphic variants of the 11beta-hydroxysteroid dehydrogenase type 1 (11ßHSD1) gene; v) assess cortisol sensitivity, expressed by the polymorphisms of the glucocorticoid receptor (GR) gene from DNA isolated from peripheral blood; vi) assess beta-2 adrenergic activity, regulated by the polymorphism (rs1800544) of the beta-2 adrenergic receptor (B2AR) gene from DNA isolated from peripheral blood, which could have an impact on cortisol effect due to the multiple interactions between the sympathetic and the hypothalamic-pituitary-adrenal systems via adrenoceptors; vii) assess gut microbiome composition, using fecal samples. To avoid the confounding effect of bone-active drugs, i), ii) and iii) will not be assessed in patients on treatment with bone-active drugs, but exclusively in naïve-treatment patients or in patients not recently treated (over 12 months previously for oral bisphosphonates and teriparatide and over 24 months previously for intravenous bisphosphonates and denosumab).

The HidHyCo case finding is of utmost importance since an underlying condition of HidHyco is associated with an increased risk of osteoporosis and fragility fractures and can decrease the response to bone-active drugs. Conversely, the resolution of cortisol excess can result in the improvement of bone strength and in the reduction of fracture risk. However, HidHyCo is by definition an occult condition, until its presence is suspected on the basis of particular characteristics of the underlying disease.

Based on preliminary data, it is possible to assume that HidHyCo is present in a not negligible percentage of osteopenic/osteoporotic patients.

The investigators hypothesize a 3% HidHyCo prevalence in the osteoporotic population. The presence of osteoporosis associated with a poorly controlled hypertension and/or diabetes or with a history of cardiovascular events (osteopenia with comorbidities) or the presence of fragility fractures in the presence of not osteoporotic bone density, in an eugonadal state and/or on osteoporotic treatment with bone-active drugs may be the variables potentially associated with an increased probability of having HidHyCo.

By testing our sample of osteoporotic patients for HidHyCo, the investigators aim at obtaining information regarding the pre-test probability of a single individual of having a subtle cortisol excess and, if feasible, at developing a clinical model for the identification in outpatient osteoporosis clinics of subjects worthy of HidHyCo testing, thus avoiding a mass screening.

Moreover, the evaluation of circulating miRNAs expression profile can help to distinguish primary osteoporosis and secondary osteoporosis due to subtle cortisol excess.

From a pathophysiological point of view, the condition of HidHyCo in our patients, differently from the exogenous hypercortisolism, may represent a pure form of slight cortisol excess, without the confounding effect of the diseases for which therapeutic glucocorticoids are given. Therefore, the assessment of bone involvement in HidHyCo patients may consent to evaluate the pure role of glucocorticoid excess on bone metabolism and bone quality, as expressed for example by the markers of bone turnover and of the Wnt-ß-catenin signaling and by the REMS parameters, respectively.

In addition, the glucocorticoid secretion and sensitivity evaluation in our osteoporotic population can also consent us to study the impact of cortisol peripheral activation and of the polymorphisms of 11ßHSD1, GR and B2AR genes in modulating the skeletal sensitivity and damage to the subtle cortisol excess.

If the importance of these parameters for bone health was confirmed, it would be possible to personalize the clinical workup on the basis of the individual risk of fracture and to try to counteract in selected patients the adverse effects of the relatively increased cortisol secretion with the 11ßHSD1 inhibitors. Indeed, some studies showed that the inhibition of the 11ßHSD1 may protect bone against the deleterious effects of glucocorticoids.

Finally, investigators will obtain information on whether or not microbiome composition differs between osteoporotic patients with and without HydHyCo. This information could suggest new pathophysiological mechanisms underlying the relationship between cortisol excess and bone fragility.

If there were interactions between these factors (microbiome and cortisol milieu) on the clinical outcomes of bone fragility, investigators might suggest the gut as a novel therapeutic target for preventing the adverse systemic effects of cortisol excess, as suggested by experimental observations. Overall, information from this study will make possible to unmask the presence of HidHyCo in patients evaluated for osteoporosis and/or bone fragility and to personalize the clinical management of these patients, in relation to the genetic background, the GC sensitivity and the microbiome composition

ELIGIBILITY:
Inclusion Criteria (one of the following):

* presence of osteoporosis (i.e. lumbar and/or femoral BMD T-score < -2.5 and/or Z-score < -2.0 and/or fragility fracture of hip, spine, wrist, humerus, malleolus or ribs);
* presence of osteopenia (i.e. lumbar and/or femoral BMD T-score between -1.0 and -2.5) in addition to hypertension treated with at least 2 drugs or not well controlled hypertension (sustained blood pressure above 150/100 mmHg) and/or diabetes and/or to a history of cardiovascular events (such as deep vein thrombosis, coronary heart disease, myocardial infarction, stroke).

Exclusion Criteria:

* pregnancy/breastfeeding, sleep apnea, prepuberal onset of hypertension, hormonal hypersecreting adrenal mass,signs/symptoms of hypercortisolism;
* already known secondary osteoporosis with the exception of hypercalciuria;
* drugs influencing the bone metabolism with the exception of diuretics, anti-diabetics and anticoagulants;
* conditions associated with increased hypothalamic-pituitary-adrenal (HPA) axis activity, severe autoimmune/rheumatologic and hematologic diseases, alcoholism, chronic kidney disease (glomerular filtration rate <60 ml/min);
* drugs influencing the HPA axis activity or the dexamethasone metabolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred to our outpatients clinics for osteoporosis
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-10-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hidden hypercortisolism in osteoporosis | 18 months
  To evaluate the prevalence of hidden hypercortisolism in patients with osteoporosis or osteopenia plus the comorbidities possibly associated with cortisol excess.
Statistical comparison of the clinical and biochemical characteristics of osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo to identify the characteristics predictive of the presence of HidHyCo in osteoporosis | 18 months
  The patients with HidHyCo (Patient Group) and those without HidHyCo (Control Group) will be compared as far as the following independent variables (taken as single variable or in combination) is concerned: i) lumbar and/or femoral BMD; ii) presence of fragility fracture; iii) presence of hypertension treated with at least 2 drugs or of not well controlled hypertension, iv) presence of diabetes; v) number of anti-hypertensive and/or antidiabetic drugs; vi) presence of a history of cardiovascular events ; vii) biochemical parameters.
  The investigators will evaluate if one or more independent variables will be associated with the presence of HidHyCo after adjusting for confounding factors. The sensitivity and specificity of the independent variables (singularly taken or in combination), which will be found to be different between the two groups in predicting the presence of HidHyCo, will be calculated.

SECONDARY OUTCOMES:
Further investigation of bone turnover in HidHyCo patients, as assessed by serum osteocalcin, CrossLaps, bone alkaline phosphatase and amino-terminal propeptide of type 1 procollagen (P1NP) and additional new potential serum markers of bone status. | 24 months
  In patients with HidHyCo and in age-, sex- and BMI-matched patients without HidHyCo investigators will assess bone turnover by measuring serum osteocalcin, CrossLaps, bone alkaline phosphatase and amino-terminal propeptide of type 1 procollagen (P1NP) and additional new potential serum markers of bone status, such as those involved in the Wnt-ßcatenin signaling (e.g. sclerostin, DKK-1 and ß-catenin levels) using commercially available kits.
Further investigation of bone quality as assessed by Radiofrequency Echographic Multi Spectrometry (REMS) | 24 months
  Radiofrequency Echographic Multi Spectrometry (REMS), a non-ionizing skeleton technique performed employing a new dedicated echographic device (EchoStation, Echolight Spa, Lecce, Italy) will be performed to further investigate bone characteristics that are not included in DXA-measured bone mineral density.
Characterization of HidHyco patients from a molecular and genetic point of view by the determination of circulating microRNAs, peripheral glucocorticoid activity and the polymorphic variants of the 11ßHSD1, GR and B2AR gene. | 24 months
  To characterize HidHyco patients from a molecular and genetic point of view investigators will assess the circulating microRNAs (i.e. small non coding single-stranded RNAs that have emerged as important post transcriptional regulators of gene expression) expression profile, the cortisol peripheral activation, as expressed by the 24-hour urinary free cortisol/free cortisone ratio, measured by liquid chromatography-tandem mass spectrometry and its relationship with the polymorphic variants of the 11beta-hydroxysteroid dehydrogenase type 1 (11ßHSD1) gene, the cortisol sensitivity, expressed by the polymorphisms of the glucocorticoid receptor (GR) gene from DNA isolated from peripheral blood, the beta-2 adrenergic activity, regulated by the polymorphism (rs1800544) of the beta-2 adrenergic receptor (B2AR) gene from DNA isolated from peripheral blood.
Assessment of gut microbiome composition by the analysis of fecal samples | 24 months
  To determine the gut microbiome composition in HidHyCo patients for the identification of the potential role of the gut microbiome in the determination of the negative effects of endogenous subtle cortisol excess on bone health.

CONTACTS AND LOCATIONS:
Overall Officials: Iacopo Chiodini, Professor, Principal Investigator — ASST Ospedale Niguarda, Milan, Italy
Locations (5):
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico "G. Rodolico-San Marco", Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Auxologico Italiano IRCCS, Milan
  - Ospedale "Casa Sollievo della Sofferenza" IRCCS, San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria Senese, Siena